CLINICAL TRIAL: NCT07172100
Title: Effect of Papaya Leaf Extract on Thrombocytopenia in Children With Dengue Fever at a Tertiary Care Center in Karachi
Brief Title: To Assess the Efficacy of Carica Papaya Leaf Extract in Improving Platelet Counts Among Pediatric Patients With Dengue-associated Thrombocytopenia
Acronym: papaya leaf
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Ziauddin Hospital (Other)
Responsible Party: Principal Investigator, Guzel Maxood, Principal Investigator, Ziauddin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6600223GMPED
Record Dates: First submitted 2025-08-20; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Dengue Fever; Papaya Leaf Extract; Pediatric Patients
Keywords: effect of papaya leaf extract; dengue fever; platelet count
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carica Papaya Leaf Extract Group (Experimental): Participants in this arm will receive oral Carica papaya leaf extract syrup (10 mL containing 1000 mg of extract), administered three times daily for 3 days, along with standard supportive care for dengue fever. Standard therapy includes hydration, antipyretics, and monitoring per hospital protocol.
  Interventions: Drug: Carica Papaya Leaf Extract Group
- Standard Therapy Group (Active Comparator): Participants in this arm will receive standard supportive treatment for dengue fever, including antipyretics, fluids, and monitoring as per institutional protocol. No Carica papaya leaf extract will be administered.
  Interventions: Other: standard treatment

INTERVENTIONS:
Drug: Carica Papaya Leaf Extract Group — Carica papaya leaf extract syrup will be administered orally at a dose of 10 mL three times daily (TID) for a total of 3 days. Each 10 mL dose contains 1000 mg of papaya leaf extract. This intervention will be given in addition to standard supportive therapy for dengue fever
  Arms: Carica Papaya Leaf Extract Group
Other: standard treatment — patients in this group will receive only the standard treatment for dengue fever
  Arms: Standard Therapy Group

SUMMARY:
The goal of this clinical trial is to evaluate whether Carica papaya leaf extract (CPLE) can improve platelet counts in children aged 2 to 12 years diagnosed with dengue fever and thrombocytopenia. The main questions it aims to answer are:

Does Carica papaya leaf extract significantly increase platelet counts compared to standard supportive therapy alone?

Does the use of Carica papaya leaf extract reduce the need for platelet transfusion or PICU admission?

Researchers will compare the group receiving CPLE plus standard therapy to the group receiving standard therapy alone to see if CPLE leads to improved platelet recovery and better clinical outcomes.

Participants will:

Be randomly assigned to receive either standard care or standard care plus Carica papaya leaf extract syrup (10 mL orally, three times daily for 3 days)

Undergo blood testing on Day 1 and Day 3 to assess platelet count, hemoglobin, WBC, and packed cell volume

Be monitored for clinical outcomes including need for transfusion and admission to the Pediatric Intensive Care Unit (PICU)

DETAILED DESCRIPTION:
Dengue fever is a mosquito-borne viral illness that continues to pose a significant health threat in tropical and subtropical regions, including Pakistan. One of the common hematological complications of dengue infection is thrombocytopenia (a low platelet count), which can lead to bleeding, requiring hospitalization, intensive care, or platelet transfusions. Currently, there is no specific antiviral treatment for dengue; management remains largely supportive.

Carica papaya leaf extract (CPLE) has shown potential as an adjunct therapy due to its proposed thrombopoietic, anti-inflammatory, and antiviral properties. Previous studies, primarily conducted in other countries, have suggested that CPLE may aid in increasing platelet counts in patients with dengue fever. However, limited data exists regarding its efficacy in pediatric populations within Pakistan.

This randomized controlled trial will be conducted to evaluate the efficacy of oral Carica papaya leaf extract in improving platelet counts in children with dengue-associated thrombocytopenia. The study will be carried out at the Department of Pediatrics, Ziauddin Hospital, Clifton Campus, Karachi, over a period of three months.

Participants will be randomly assigned into two groups:

Intervention group (n=55): Will receive 10 mL of Carica papaya leaf extract syrup orally three times daily (each 10 mL dose containing 1000 mg of extract) along with standard supportive therapy.

Control group (n=52): Will receive standard supportive therapy alone.

The primary objective of the study is to assess whether CPLE significantly increases platelet counts from Day 1 to Day 3 compared to standard therapy alone. Secondary objectives include evaluating changes in hemoglobin levels, white blood cell (WBC) count, packed cell volume (PCV), need for platelet transfusion, and admissions to the Pediatric Intensive Care Unit (PICU).

Baseline demographics (age, gender, height, and weight) will be recorded. Laboratory tests including complete blood count will be conducted on Day 1 and Day 3. Data will be analyzed to determine whether CPLE leads to meaningful clinical improvements beyond standard care.

This study is expected to contribute important local data regarding the use of CPLE in pediatric dengue cases. If effective, this herbal adjunct could offer a low-cost, accessible therapeutic option. However, if no benefit is observed, the findings will help guide clinical practice away from potentially unnecessary interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dengue fever
* Patients from age 2 till 2 years of age

Exclusion Criteria:

* Patients hypersensitive to papaya leaf extract
* Patients with bleeding disorder

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Platelet Count from Day 1 to Day 3 | Baseline (Day 1) and Day 3
  To evaluate the effectiveness of Carica papaya leaf extract in increasing platelet count in pediatric patients with dengue-associated thrombocytopenia

CONTACTS AND LOCATIONS:
Locations (1):
- Guzel Maxood, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: Yes